CLINICAL TRIAL: NCT01067092
Title: MATCH: The Mexican-American Trial of Community Health Workers
Acronym: MATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven K. Rothschild, MD, Associate Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01DK061289 (NIH); R01DK061289 (NIH)
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community Health Worker Intervention (Experimental): A Community Health Worker makes 36 home visits to the person with diabetes over a two year period, providing diabetes education and self-management skills training. The curriculum covers recommended diabetes self-management behaviors including glucose self-monitoring, responding to abnormal blood glucose levels, working effectively with health care providers, medication adherence, foot care, daily physical activity, and reducing fat content of diet. CHWs also deliver training in behavioral skills of self-monitoring, environmental restructuring, engagement of social support, stress management, and problem-solving skills to facilitate the self-management activities.
  Interventions: Behavioral: Community Health Worker Intervention
- Educational Newsletter (Active Comparator): Diabetes education and self-management skills training delivered via 36 bilingual diabetes education newsletters over a 2 year period. The newsletters cover recommended diabetes self-management behaviors including glucose self-monitoring, responding to abnormal blood glucose levels, working effectively with health care providers, medication adherence, foot care, daily physical activity, and reducing fat content of diet. The newsletters also describe behavioral skills of self-monitoring, environmental restructuring, engagement of social support, stress management, and problem-solving skills to facilitate the self-management activities.
  Interventions: Behavioral: Educational Newsletter

INTERVENTIONS:
Behavioral: Community Health Worker Intervention — A Community Health Worker makes 36 home visits to the person with diabetes over a two year period, providing diabetes education and self-management skills training. The curriculum covers recommended diabetes self-management behaviors including glucose self-monitoring, responding to abnormal blood glucose levels, working effectively with health care providers, medication adherence, foot care, daily physical activity, and reducing fat content of diet. CHWs also deliver training in behavioral skills of self-monitoring, environmental restructuring, engagement of social support, stress management, and problem-solving skills to facilitate the self-management activities.
  Other Names: Promotora; Promotora de Salud
  Arms: Community Health Worker Intervention
Behavioral: Educational Newsletter — Diabetes education and self-management skills training delivered via 36 bilingual diabetes education newsletters over a 2 year period. The newsletters cover recommended diabetes self-management behaviors including glucose self-monitoring, responding to abnormal blood glucose levels, working effectively with health care providers, medication adherence, foot care, daily physical activity, and reducing fat content of diet. The newsletters also describe behavioral skills of self-monitoring, environmental restructuring, engagement of social support, stress management, and problem-solving skills to facilitate the self-management activities.
  Arms: Educational Newsletter

SUMMARY:
The MATCH study (Mexican-American Trial of Community Health Workers) tests the hypothesis that the use of indigenous Community Health Workers (CHWs), recruited from the target community and trained to provide culturally appropriate diabetes education, can promote pro-active self-management among inner-city dwelling Mexican-Americans with Type 2 diabetes mellitus. The study aims are to demonstrate that a CHW, compared to an attention control, will: 1) result in improvement in short term physiologic outcomes (Hemoglobin A1c levels and blood pressure), and 2) result in increased frequency of self-management behaviors (daily self blood-glucose monitoring, medication adherence, adherence to diet and physical activity recommendations). The study design is a single site, partially blinded, randomized controlled trial of 144 patients with Type 2 diabetes mellitus.

Eligibility criteria include a diagnosis of Type 2 diabetes, residence in target community areas in the Chicago area, and Mexican or Mexican-American ethnic heritage. Participants are randomized to either an experimental group receiving 36 home visits over a two year period in which a CHW delivered diabetes education and self-management skills training, or to an attention control consisting of 36 bilingual diabetes education newsletters covering the same curriculum as the CHWs. The curriculum covers recommended diabetes self-management behaviors including glucose self-monitoring, responding to abnormal blood glucose levels, working effectively with health care providers, medication adherence, foot care, daily physical activity, and reducing fat content of diet. CHWs also deliver training in behavioral skills of self-monitoring, environmental restructuring, engagement of social support, stress management, and problem-solving skills to facilitate the self-management activities. Consistent delivery of the CHW intervention is documented by audiotapes and Documentation of Intervention worksheets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Taking at one oral medication daily to control diabetes
* Self-identified as Mexican or Mexican-American
* Resident in target community within Chicago, Berwyn, or Cicero, Illinois.

Exclusion Criteria:

* Diabetes controlled with diet or insulin only
* Advanced end-organ complications, including: end-stage renal disease, stroke with paresis, Congestive Heart Failure (NYHA class 3 or 4), or other major end-organ complication of diabetes
* Receiving treatment for a major psychiatric disorder (i.e. schizophrenia)
* Are unable to understand and give informed consent in either English or Spanish
* Live in a household with someone who is already a randomized study participant or know of family members who are already study participants.
* Have lived in Mexico for more than four months in the past two years, or are anticipating extended travel to Mexico in the next year.
* Are under the age of 18

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2005-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 2 years
% of persons with blood pressure less than 130/80 | 2 years

SECONDARY OUTCOMES:
Medication adherence | 2 years
Daily self-blood glucose monitoring | 2 years
Summary of Diabetes Self-Care Activities | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Swider SM, Martin M, Lynas C, Rothschild S. Project MATCH: training for a promotora intervention. Diabetes Educ. 2010 Jan-Feb;36(1):98-108. doi: 10.1177/0145721709352381. Epub 2009 Dec 11. PMID 20008279
- [Background] Martin MA, Swider SM, Olinger T, Avery E, Lynas CM, Carlson K, Rothschild SK. Recruitment of Mexican American adults for an intensive diabetes intervention trial. Ethn Dis. 2011 Winter;21(1):7-12. PMID 21462723